CLINICAL TRIAL: NCT07258355
Title: Occupation-Based Multicomponent Intervention to Reduce Fall Risk in Older Adults Living in a Community With a History of Falls: A Prospective Quasi-Experimental Study
Brief Title: Occupation-Based Multicomponent Intervention to Reduce Fall Risk in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Medine Nur Özata Değerli, Research Assistant, Occupational Therapist, PhD Candidate, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4fba1e62c6f1465b
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Geriatric; Fall; Cognition; Balance; Occupational Therapy
Keywords: Occupational therapy; Fall prevention; Older adults; Occupation-based intervention; Balance and gait

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occupation-Based Multi-Component Intervention (Experimental)
  Interventions: Behavioral: Occupation-Based Multi-Component Intervention

INTERVENTIONS:
Behavioral: Occupation-Based Multi-Component Intervention — Occupation-Based Multi-Component Intervention

SUMMARY:
This study aims to examine the effects of an occupation-based, multicomponent occupational therapy intervention on older adults aged 65 years and above with a history of falls living in the community. The intervention consists of 12 individualized sessions designed around the participants' meaningful occupations. It incorporates balance and gait training, environmental modifications, behavioral strategies, and safety-enhancing activities within a holistic framework. The sample will include 40 older adults who have experienced at least one fall in the past year. Data will be collected using the Canadian Occupational Performance Measure (COPM), Tinetti Balance and Gait Test, Timed Up and Go Test (TUG), and Mini-Mental State Examination (MMSE). Pre- and post-intervention measurements will be compared to evaluate the program's effects on occupational performance, satisfaction, balance, and gait functions. The study is expected to provide valuable evidence on the effectiveness of occupation-based approaches in fall prevention interventions for older adults.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of a 12-session occupation-based, multicomponent occupational therapy intervention for older adults aged 65 years and above who have a history of falls. Falls are common in this population and are influenced by a combination of physical, behavioral, and environmental factors. Occupational therapy interventions that integrate balance training, environmental modification, and activity-based strategies may support safer participation in daily occupations. The intervention in this study is individualized and structured around the meaningful occupations identified by participants through the Canadian Occupational Performance Measure (COPM). The program includes components such as balance and gait training during daily activities, safety education, environmental adaptations, and behavioral strategies to reduce fall risk. Sessions are conducted individually in a face-to-face format and include both clinic-based and real-environment activities. Participants will complete standardized assessments before and after the intervention, including measures of occupational performance, satisfaction, balance, and functional mobility. The results will contribute to the understanding of how occupation-based multicomponent interventions support fall prevention and functional independence in community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria

History of at least one fall within the last 6 months

Age 65 years or older

Exclusion Criteria

Presence of a primary neurological condition that could contribute to falls (e.g., stroke, Parkinson's disease)

Presence of an orthopedic condition that could contribute to falls (e.g., extremity fractures, osteoarthritis, limb length discrepancy)

Presence of a psychiatric condition that could contribute to falls

History of any surgical operation involving the extremities

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination | 12 week
  It is one of the most widely used cognitive screening tools. It consists of five main sections-orientation, immediate recall, attention and calculation, delayed recall, and language-covering a total of 11 items. Scores range from 0 to 30, with higher scores indicating better cognitive functioning. The Turkish validity and reliability study has been conducted, and a cut-off score of 23/24 is commonly recommended for the Turkish population.
Canada Occupational Performance Measurement | 12 week
  It will be used to identify the daily occupations that older adults want to do, need to do, or are expected to do, as well as to determine which of these occupations are affected by current difficulties. The COPM allows individuals to identify activities within the categories of self-care, leisure, and productivity. From these, five priority activities are selected, and the individual rates both their occupational performance and satisfaction for each activity on a scale from 1 to 10. Higher scores indicate better performance and greater satisfaction. The scores for performance and satisfaction are summed and divided by the number of selected activities to obtain mean performance and satisfaction scores.
Tinetti Balance and Gait Test | 12 week
  The Tinetti scale evaluates an individual's balance and gait abilities through two components: balance (9 items) and gait (7 items), each reflecting movements commonly performed during daily activities. Each item is scored from 0 to 2, where 2 indicates correct and safe performance, 1 indicates performance with adaptations, and 0 indicates inability to perform the movement. The balance items generate a balance score, the gait items generate a gait score, and their sum constitutes the total score, which indicates fall risk. A total score of 18 or below reflects a high fall risk, 19-24 indicates a moderate risk, and 25 or above indicates a low fall risk. The scale is widely used and considered valid and reliable for older adults.
Timed Up and Go test | 12 week
  The TUG test assesses dynamic balance, fall risk, and functional mobility in older adults. During the test, the individual is asked to stand up from a chair, walk a distance of three meters, turn around, walk back to the chair, and sit down. The total time to complete the sequence is recorded as the test result.
  A duration longer than 12 seconds indicates decreased functional performance during daily activities and a higher risk of falling. The test is simple, quick to administer, and widely used in geriatric assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Universitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leland NE, Elliott SJ, O'Malley L, Murphy SL. Occupational therapy in fall prevention: current evidence and future directions. Am J Occup Ther. 2012 Mar-Apr;66(2):149-60. doi: 10.5014/ajot.2012.002733. PMID 22394524
- [Result] Kim M, Shin E, Kim S, Sok S. The Effectiveness of Multicomponent Intervention on Daily Functioning among the Community-Dwelling Elderly: A Systematic Review. Int J Environ Res Public Health. 2022 Jun 18;19(12):7483. doi: 10.3390/ijerph19127483. PMID 35742730
- [Result] James SL, Lucchesi LR, Bisignano C, Castle CD, Dingels ZV, Fox JT, Hamilton EB, Henry NJ, Krohn KJ, Liu Z, McCracken D, Nixon MR, Roberts NLS, Sylte DO, Adsuar JC, Arora A, Briggs AM, Collado-Mateo D, Cooper C, Dandona L, Dandona R, Ellingsen CL, Fereshtehnejad SM, Gill TK, Haagsma JA, Hendrie D, Jurisson M, Kumar GA, Lopez AD, Miazgowski T, Miller TR, Mini GK, Mirrakhimov EM, Mohamadi E, Olivares PR, Rahim F, Riera LS, Villafaina S, Yano Y, Hay SI, Lim SS, Mokdad AH, Naghavi M, Murray CJL. The global burden of falls: global, regional and national estimates of morbidity and mortality from the Global Burden of Disease Study 2017. Inj Prev. 2020 Oct;26(Supp 1):i3-i11. doi: 10.1136/injuryprev-2019-043286. Epub 2020 Jan 15. PMID 31941758
- [Result] Gillespie LD, Gillespie WJ, Robertson MC, Lamb SE, Cumming RG, Rowe BH. Interventions for preventing falls in elderly people. Cochrane Database Syst Rev. 2003;(4):CD000340. doi: 10.1002/14651858.CD000340. PMID 14583918
- [Result] Fernandez-Arguelles EL, Rodriguez-Mansilla J, Antunez LE, Garrido-Ardila EM, Munoz RP. Effects of dancing on the risk of falling related factors of healthy older adults: a systematic review. Arch Gerontol Geriatr. 2015 Jan-Feb;60(1):1-8. doi: 10.1016/j.archger.2014.10.003. Epub 2014 Nov 6. PMID 25456888
- [Result] Altuntas O, Degerli MNO, Temizkan E, Ekici G. Psychometric properties of the Canadian occupational performance measure in older individuals. Turk J Med Sci. 2023 Nov 28;54(1):338-347. doi: 10.55730/1300-0144.5796. eCollection 2024. PMID 38812638